CLINICAL TRIAL: NCT07243574
Title: Night Owl Sleep Study: The Effect of Sleep on Fecal Microbiota
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IFF-NO-001
Record Dates: First submitted 2025-09-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): Cohort 1 are participants who have insufficient sleep at baseline; this cohort will be assigned to spend 1.5 hours more in bed per night.
  Interventions: Behavioral: Increase sleep by 90 minutes
- Cohort 2 (Active Comparator): Cohort 2 are participants who have sufficient sleep at baseline; this cohort will be assigned to spend 1.5 hours less in bed per night.
  Interventions: Behavioral: Decrease sleep by 90 minutes

INTERVENTIONS:
Behavioral: Increase sleep by 90 minutes — For 14 days, participants will increase their nightly sleep by 90 minutes.
  Arms: Cohort 1
Behavioral: Decrease sleep by 90 minutes — For 14 days, participants will decrease their nightly sleep by 90 minutes.
  Arms: Cohort 2

SUMMARY:
The goal of this clinical trial is to assess differences in the fecal microbiota and metabolome associated with insufficient and sufficient sleep, and to evaluate the response and recovery of the microbiota to changes in participant sleep profiles.

Researchers will compare the effect of sleep intervention on both insufficient and sufficient sleepers to identify differences in fecal microbiota structure and function between cohorts during habitual sleep and during the sleep alteration intervention period..

Participants will be assigned to one of two cohorts based on their current sleep habits. Cohort 1 are participants who have insufficient sleep at baseline; this cohort will be assigned to spend 1.5 hours more in bed per night. Cohort 2 are participants who have sufficient sleep at baseline; this cohort will be assigned to spend 1.5 hours less in bed per night. The sleep intervention lasts for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 20 - 40 years of age (inclusive).
2. Currently employed and have been employed for at least 6 months, at least 30 hours a week.
3. Consistent work schedule during daytime hours with weekends off.
4. BMI 18.5 - 30 kg/m2 (inclusive).
5. Good physical and mental health as established by self-reported medical history.
6. Willingness to maintain and record their general habits, eating, and activity/exercise pattern for the study period.
7. Willingness to maintain and record the same time in bed they have during the workdays throughout the habitual workday sleep period
8. Able to alter sleeping time during the study intervention period as instructed.
9. Willingness to maintain typical sleep hygiene patterns (e.g. sleep location, temperature, environment).
10. Willingness to maintain their current pattern of alcohol consumption for the duration of the study.
11. Willing and able to participate fully in all aspects of the study and complete all study procedures, including providing signed informed consent.
12. Completes all study procedures during the 14-day screening period to be eligible for the cohort specifi c criteria based on the sleep data collected during screening period.
13. Has regular bowel habits and would be able to consistently pass stool in the morning every day.
14. Pittsburgh Sleep Quality Index (PSQI) score ≤7.

Cohort 1 (Insufficient Sleep)

Participants must meet all general inclusion criteria PLUS:

1. Sleep, on average, 5-6 hours per night on workdays, verified via participant self-report during the screening period.
2. Report extending their sleep during free (non-workday) days for an average of more than 75 minutes, verified via participant self-report during the screening period.
3. Report feeling sleepy and regularly desiring to nap during the daytime, with a score of ≥ 10 on the ESS evaluated during the screening period.
4. Average KSS Score of 6-10 on workdays during the screening period.

Cohort 2 (Sufficient Sleep)

Participants must meet all general inclusion criteria PLUS:

1. Sleep, on average, 7-8 hours per night on workdays, verifi ed via participant self-report during the screening period.
2. Do not extend sleep on free (non-workday) days by more than 45 minutes, verifi ed via participant self-report during the screening period.
3. No consistent sleep deprivation or need for nap, with a score of ≤9 on the ESS evaluated during the screening period.
4. Average KSS Score of 1-5 on workdays during screening period

Exclusion Criteria:

1. Any current diagnosed or self-reported sleep or gastrointestinal disorder, including sleep apnea, habitual snoring, insomnia, narcolepsy, parasomnias, Crohn's disease, ulcerative colitis, celiac disease, IBS, or functional bowel disorder or chronic heart burn.
2. Tendency to wake up during the night or be woken up by a partner, pet, or child(ren).
3. Chronic conditions requiring medication that, in the investigator's opinion, may affect the participants' microbiome or sleep.
4. Neurodegenerative diseases (including multiple sclerosis, Parkinson's disease, Alzheimer's disease, dementia).
5. Recent history (past year) of alcohol or drug abuse or dependence, including consistent recreational substance use such as marijuana.
6. Binge drinking behavior, defined as 4 or more alcoholic drinks for women or 5 or more alcoholic drinks for men in one sitting, within the past 3 months.
7. Diagnosed neuropsychiatric disorders or symptoms possibly affecting sleep (generalized anxiety disorder (GAD), major depressive disorder (MDD), bipolar disorder, schizophrenia)
8. Use of medications or dietary supplements to initiate or maintain sleep within 4 weeks prior to screening, including, but not limited to, melatonin, diphenhydramine (Benadryl), magnesium, sedative or hypnotic medications (i.e. zopiclone, zolpidem), and benzodiazepines.
9. Use of medications with clinically significant effects on sleep, including, but not limited to, SSRIs, beta agonists, sulphonylureas, beta antagonists, opiate analgesics, alpha antagonists, stimulants, and glucocorticoids within the past 3 months.
10. Any use of systemic antibiotics in the past 3 months. Topical or targeted antibiotic use (eye drop, ear drop) are allowed.
11. Any use of probiotic supplements in the past 2 weeks.
12. Any use of proton pump inhibitors (PPIs) in the past 2 weeks.
13. Pregnant or breastfeeding or planning to become pregnant.
14. Personal life situation causing stress or challenges in sleep (eg. caretaker required to wake up during sleep, major change in personal life).
15. Planned overnight or cross time zone travel during the study.
16. Females experiencing perimenopausal or menopausal symptoms, or those who have been diagnosed as perimenopausal or menopausal by a physician.
17. Any diagnosed condition or undiagnosed symptom which disrupts sleep, including, but not limited to, hyperthyroidism, night sweats, restless legs, or poorly controlled allergic rhinitis.
18. Extreme chronotypes; those that regularly go to sleep prior to 08:00 pm or after 2:30 am.
19. Varying work schedule, including shift workers who work late or overnight shifts or rotating schedules.
20. Any other personal or medical condition that the investigator believes may bias or confound the results.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Differences in the fecal microbiota of individuals with sufficient and insufficient sleep. | From Day 1 to Day 28
  Measure changes in microbial abundance and diversity from baseline to the end of the study in those individuals who have sufficient sleep compared to those with insufficient sleep. This is comparing the sufficient sleep group to the insufficient sleep group across all study periods.
To evaluate the response of the microbiota to changes in participant sleep duration. | From Day 1 to Day 28
  Measure changes in gut microbiota within the individual during times of sufficient sleep compared to when they are getting insufficient sleep.This is measuring the change within individual participants before the intervention and after.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Global Life Research Network, Miami, Florida
  - Lindus Health, Boston, Massachusetts
  - AccuMed, Garden City, New York

IPD SHARING:
Plan to Share IPD: No